CLINICAL TRIAL: NCT06809296
Title: Evaluating the Effects of Acute Exposure to Cold and Heat on Appetite: Impact of Serving Food Temperature (Hot and Cold Meals)
Brief Title: Assessment of the Effects of Acute Exposure to Cold and Heat on Appetite
Acronym: TEMPCA2
Status: Not yet recruiting | Type: Observational
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Collaborators: Institut de recherche biomédicale des armées (IRBA), Bretigny sur Orge, France (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2024PPRC09; 2024-A02285-42 (Other: IDRCB)
Record Dates: First submitted 2025-01-22; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Appetite
Keywords: Appetite; food intake; Thermal exposure; Cold; Heat; Energy intake
MeSH Terms: conditions — Common Cold

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Warm Meal (WM): This group will receive an ad libitum warm meal at 01:00pm after 4h30 of exposure to threee different thermal environments
- Cold Meal: This group will receive an ad libitum cold meal at 01:00pm after 4h30 of exposure to threee different thermal environments

SUMMARY:
Military personnel and athletes have a very high energy expenditure, which is increased during certain key periods (intense training, competition and missions). Compensating for this expenditure through adequate energy intake can be complicated by physiological ingestive limits and logistical and organizational constraints (number of meals, food availability), leading these populations to regularly find themselves in an energy deficit situation (intake below requirements). If this situation persists, it could impair physical and cognitive performance, as well as major physiological functions. Among the many constraints to which military personnel and athletes are subjected (stress, sleep deprivation, travel, etc.) that can increase the risk of energy deficiency, the impact of thermal environmental constraints is very imperfectly known. Seasonal impact and travel to countries with very different thermal environments from temperate countries can lead these populations to work in cold and hot conditions for long periods.

Understanding how exposure to hot and cold alters appetite and energy intake is therefore of the high importance. Our previous "TEMPCA" study highlighted a modulation of preferences for warm or cold foods depending on the exposure environment. By being able to adapt their food intake to these preferences, subjects were able to maintain a decent energy intake.

The primary objective of this study is to determine the effect of the temperature of the food served (hot or cold) on changes in food intake during acute exposure to hot and cold. We hypothesized that adapting the temperature of the food served according to the exposure environment (hot in a cold environment and cold in a hot environment) would enable adequate levels of energy intake.

Secondary objectives are to determine the influence of the environment on the levels of interstitial glucose during the preprandial period and to investigate the impact of thermal exposure (modulation of core temperature) on the modulation of quantities consumed and energy produced by digestion (postprandial thermogenesis). Forty participants (between 18 and 40 yo, male or female, active, lean, and healthy) will carry out 3 experimental sessions in which only the thermal environment will differ: cold condition (15°C), neutral condition (25°C) and warm condition (35°C). They will be divided into two groups, the first of which will be offered a cold meal during the three sessions (Cold Meal - CM) and the second a warm meal during the three sessions (Warm Meal - WM). They will all wear the same outfit designed to be offer perfect thermal comfort at 25 °C.

Briefly, each session will start at 8:30am after eating a standardized breakfast. Body mass and ad libitum water intake will be frequently monitored to identify possible dehydration. Thermal comfort and sensation and subjective appetite will be regularly assessed using visual analog scale.

From 11:00am to 01:00pm, all participants will be isolated and all temporal cues will be removed. At 01:00pm, an ad libitum meal (warm or cold) will be served in large quantities. The dishes will be weighed before and after the meal to assess energy intake. Before and after the meal, resting metabolism will be measured during 30 min in a supine position using indirect calorimetry and food preferences for high-fat/low-fat, savory/sweet, warm/cold foods, and fluid/solid foods will be assessed using the Leeds Food Preference Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Active (>3 h/w of physical activites)
* Affiliated to the social security
* Usual breakfast eaters

Exclusion Criteria:

* Unusual or irregular meal pattern
* Too high dietary restrictive profile assessed by the TFEQ-21
* Bad sleepers (< 6h/night)
* Presenting a metabolic condition
* BMI lower than 18 or higher than 30
* Chronic medication (at the exception of the contraceptive pills)
* Regular smoker (more than 2 cigarettes per day)
* Regular alcohol consumer (more then 1 glass per day)
* Vegetarian
* Following a confessional diet (hallal, casher)
* Do not speak fluently French

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Active, young, lean, healthy individuals and presenting normal diet and sleep patterns.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Energy intake | From date of the first experimental session until the last experimental session
  Energy intake measured during the test ad libitum meal served at 01:00pm.
Subjective appetite | From date of the first experimental session until the last experimental session
  Hunger, desire to eat, prospective consumption, gastric fullness, and thirst feelings will be assessed using 10-cm visual analog scales each hour from the begininng (8:30 am) to the end of the exposure (03:00pm)
Food preferences | From date of the first experimental session until the last experimental session
  Food preferences for high-fat/low-fat, sweet/savory foods and for warm/cold and fluid/solid foods will be assessed using the Leeds Food Preference Questionnaire at 12:30am and 01:30pm

SECONDARY OUTCOMES:
Rectal temperature | From date of the first experimental session until the last experimental session
  Using a rectal probe continuously during the three thermal exposures
Skin temperature | From date of the first experimental session until the last experimental session
  Using 4 thermobuttons on 4 different sites (chest, arm, thigh and back) continuously during the three thermal exposures
Thermal sensation and comfort | From date of the first experimental session until the last experimental session
  Using visual analog scales each hour from the begininng (8:30 am) to the end of the exposure (03:00pm)
Levels of interstitial glucose | From date of the first experimental session until the last experimental session
  Using a Freestyle Libre 2 (continuous glucose monitoring system) with a 5-min sample rate continuously during the three thermal exposures
Resting energy metabolism | From date of the first experimental session until the last experimental session
  Using the Q-NRJ (Cosmed) during a 30-min measurement in a supine position 60 minutes before the meal (12:00 am) and 60 minutes after the meal (02:00 pm)

CONTACTS AND LOCATIONS:
Overall Officials: Keyne Charlot, PhD, Principal Investigator — Institut de Recherche Biomédical des Armées

IPD SHARING:
Plan to Share IPD: Yes
All data and will be make available for other researchers on request.
Supporting Information: Study Protocol, SAP
Time Frame: IPD will be available when an article will be published.
Access Criteria: Any researcher that will make a demand using e-mail address of the corresponfing author. They will have access to individual and mean data and the explanation of the gathered outcomes.

REFERENCES:
- [Result] Tassone EC, Baker BA. Body weight and body composition changes during military training and deployment involving the use of combat rations: a systematic literature review. Br J Nutr. 2017 Mar;117(6):897-910. doi: 10.1017/S0007114517000630. PMID 28452292
- [Result] Wasse LK, King JA, Stensel DJ, Sunderland C. Effect of ambient temperature during acute aerobic exercise on short-term appetite, energy intake, and plasma acylated ghrelin in recreationally active males. Appl Physiol Nutr Metab. 2013 Aug;38(8):905-9. doi: 10.1139/apnm-2013-0008. Epub 2013 May 1. PMID 23855280
- [Result] Zakrzewski-Fruer JK, Horsfall RN, Cottrill D, Hough J. Acute exposure to a hot ambient temperature reduces energy intake but does not affect gut hormones in men during rest. Br J Nutr. 2021 Apr 28;125(8):951-959. doi: 10.1017/S0007114520002792. Epub 2020 Jul 22. PMID 32693846
- [Result] Charlot K. Negative energy balance during military training: The role of contextual limitations. Appetite. 2021 Sep 1;164:105263. doi: 10.1016/j.appet.2021.105263. Epub 2021 Apr 20. PMID 33862189
- [Result] Millet J, Siracusa J, Tardo-Dino PE, Thivel D, Koulmann N, Malgoyre A, Charlot K. Effects of Acute Heat and Cold Exposures at Rest or during Exercise on Subsequent Energy Intake: A Systematic Review and Meta-Analysis. Nutrients. 2021 Sep 28;13(10):3424. doi: 10.3390/nu13103424. PMID 34684424
- [Result] Coca M, Besancon L, Erblang M, Bourdon S, Gruel A, Lepetit B, Beauchamps V, Tavard B, Oustric P, Finlayson GS, Thivel D, Malgoyre A, Tardo-Dino PE, Bourrilhon C, Charlot K. Twenty four-hour passive heat and cold exposures did not modify energy intake and appetite but strongly modify food reward. Br J Nutr. 2024 Jul 28;132(2):209-226. doi: 10.1017/S0007114524000825. Epub 2024 Apr 18. PMID 38634266